CLINICAL TRIAL: NCT04350944
Title: FGF-23 and PTH During Hemodialysis Patients Under Consideration of Calcification Propensity - a Pilot Study
Brief Title: FGF-23 and PTH in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rainer Oberbauer, Univ.-Prof. Rainer Oberbauer, MD, PhD, Medical University of Vienna
Other Study IDs: FGF-23 and PTH during HD
Record Dates: First submitted 2020-03-22; First posted 2020-04-17 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: CKD; Hemodialysis; FGF 23; PTH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Three samples per patient and dialysis treatment will be drawn at the start, after 2 hours and at the end of dialysis. Blood samples will be collected from the dialysis machine. Blood is allowed to clot, serum and plasma will be separated by centrifugation and kept in aliquots (500µl) at -80° until further analysis.
  Parathyroid hormone (PTH), Serum calcium (sCa), phosphate (P), 25-hydroxy-vitamin D (25(OH)D) and 1,25 dihydroxy-vitamin D (1,25(OH)2D) will be determined by routine assays at the Department of Laboratory Medicine of the General Hospital of Vienna. FGF-23 will be determined by an iFGF-23 enzyme-linked immunosorbent assays (ELISA) of Biomedica and the T50-time will be measured by an nephelometer at the Calciscon Laboratory in Switzerland.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this pilot study the investigator will examine the levels of fibroblast growth factor (FGF-23) and parathyroid hormone (PTH) levels during hemodialysis therapy in 30 patients and assess the correlation between these parameters and the T-50 calcification propensity, as well as further parameters of secondary hyperparathyroidism (sHPT), like serum calcium (sCa), phosphate (P), 25-hydroxy-vitamin D (25(OH)D) and 1,25 dihydroxy-vitamin D (1,25(OH)2D).

The investigator hypothesize that FGF-23 and PTH levels are at their highest at the beginning of dialysis and decrease during the treatment.

DETAILED DESCRIPTION:
Background: The development of sHPT in hemodialysis patients is a common complication which induces an increase in calcification and atherosclerosis. Elevated FGF-23 levels are already found in early stages of chronic kidney disease (CKD) and it has been shown that high FGF-23 levels are associated with the development of cardiovascular disease and increased overall mortality.

Method: In this pilot study a total number of 30 patients on maintenance haemodialysis will be enrolled. The investigator will examine the course of FGF-23 and PTH levels during a single hemodialysis session. In addition, the T-50 time, a novel non-traditional cardiovascular risk factor as well as further parameters of sHPT, such as serum calcium (sCa), phosphate (P), 25-hydroxy-vitamin D (25(OH)D) and 1,25 dihydroxy-vitamin D (1,25(OH)2D) will be assessed.

Hypothesis and specific aims: The major end point of the study is the level of FGF-23 and PTH at three points during hemodialysis treatment. As secondary end points the T-50 calcification propensity and further parameters of sHPT, as well as the correlation between these parameters will be measured.

Hemodialysis is classified as a kidney replacement therapy and FGF-23 and PTH are partly metabolized and excreted by the kidneys. Based on this the investigator hypothesize that FGF-23 and PTH levels are at their highest at the beginning of dialysis and decrease during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* hemodialysis three times a week

Exclusion Criteria:

* Subject is currently enrolled or not yet completed at least 30 days since ending other investigational device or drug trial(s), or is receiving other investigational agent(s)
* Pregnancy
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with the study procedures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 adult patients with chronic kidney disease receiving hemodialysis treatment at the Medical University of Vienna, Department of Internal Medicine III, Division of Nephrology and Dialysis. All patients are on a thrice-weekly dialysis schedule.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Time course of FGF-23 and PTH levels during hemodialysis treatment. | 1 day
  This trial is designed to analyze the levels of fibroblast growth factor 23 and parathyroid hormone concentrations during hemodialysis treatment. Measurements will be performed at three timepoints during one single treatment session on one single treatment day. The first measurement will be performed at the beginning of dialysis (just after connecting the patient to the dialysis machine), the second after two hours of dialysis and the third at the end of the dialysis treatment (before disconnecting the patient from the machine).

SECONDARY OUTCOMES:
T-50 calcification, sHPT parameters | 1 day
  T-50 calcification propensity and further parameters of secondary hyperparathyroidism (serum calcium, phosphate and vitamin D) as well as the correlation between these parameters. Measurements will be performed at the beginning of dialysis (just after connecting the patient to the dialysis machine).

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Oberbauer, MD, PhD, Principal Investigator — Head of the department of Nephrology and Dialysyis of the MUV
Locations (1):
- Medical University of Vienna, Vienna, Austria